CLINICAL TRIAL: NCT04095871
Title: Determinants, Impact and Adherence Related to the Duration of Performing Self Catheterization on Patient Satisfaction and Quality of Life
Status: Completed | Type: Observational
Sponsor: Gérard Amarenco (Other)
Responsible Party: Sponsor-Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Organization: Pierre and Marie Curie University (Other)
Other Study IDs: GRC -- 01GREEN
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Intermittent Urethral Catheterization; Lower Urinary Tract Symptoms; Treatment Adherence; Patient Satisfaction
Keywords: Intermittent urethral catheterization; Treatment adherence and compliance; Lower urinary tract symptoms; Urinary retention; Patient satisfaction
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Treatment Adherence and Compliance; Patient Satisfaction; Urinary Retention | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients included: Patients over 18 years old performed CISC for more than 1 month, exclusive or not, are included.
  At home, patients have to complete one diary on the specific duration of a 24-hour CISC and the next day a second diary on the total duration of CISC.
  The specific time of CISC described by the timed duration from the moment when the circumstances of care are combined to carry it out : isolated place, nearby equipment.
  The total time of CISC described by the timed duration from the moment of the intention to self-catheter until the return to the initial activity.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention, patients record the time of CISC
  Other Names: no intervention

SUMMARY:
Clean Intermittent Self-Catheterization (CISC) is a procedure of regularly emptying the bladder by introducing a single-use urinary catheter through the urethra. CISC are indicated in several situations in patients with neurological pathologies but also with urological or functional disorders.

The announcement of the indication of CISC is often difficult and the acceptance of this therapy remains complicated, due to the invasive side, the dependence on a material and the time required to perform CISC.

A few studies have assessed patient satisfaction and adherence to self-catheterization through quality of life questionnaires, but none have examined the impact of this technique on daily life through the duration of CISC.

Primary aim is to evaluate the impact of time to perform CISC on patient adherence and satisfaction.

Patients over 18 years old performed CISC for more than 1 month, exclusive or not, are included.

History and treatment, age, professional activity, visuals disorders, technical aids for walking and the history of CISC with the date of initiation, the type of catheter, the carrier, the number of CISC per 24 hours, the position of realization, the use of a mirror and urethral sensitivity are recorded. Cognitive disorders, fatigue, psychological state, impact on quality of life are assessed on the day of the patient's consultation. The grip of the upper limbs is explored by Box and Block and Nine Hole Peg Test. The validated questionnaires,Intermittent Catheterization Satisfaction Questionnaire ( InCaSaQ), Intermittent Catheterization Difficulty Questionnaire (ICDQ), Intermittent Catheterization Adherence Scale (ICAS) are completed.

At home, patients have to complete one calendar on the specific duration of a 24-hour self-catheterization and the next day a second calendar on the total duration of CISC

Primary outcome is specific time of self-catheterization described by the timed duration from the moment when the circumstances of care are combined to carry it out : isolated place, nearby equipment.

Secondary outcome is total time of self-catheterization described by the timed duration from the moment of the intention to self-catheter until the return to the initial activity.

Influence of age, Expanded Disability Status Scale (EDSS), American Spinal Injury Association (ASIA), Montreal Cognitive Assessment (Moca), Fatigue Impact Scale (FIS), Box and Block and Nine Hole Peg Test, Hospital Anxiety and Depression Scale (HADS), Qualiveen Total,Intermittent Catheterization Satisfaction Questionnaire (InCaSaQ), Intermittent Catheterization Difficulty Questionnaire (ICDQ), Intermittent Catheterization Adherence Scale (ICAS) on time of self-catheterization are analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years of age perform sel-catheterization since more than 1 month (they could keep spontaneous voiding associated with CISC.

Exclusion Criteria:

* patients with an inability to comply with protocol instructions (severe cognitive disorders, language barrier, assistance with AS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients >18 years of age perform sel-catheterization since more than 1 month (they could keep spontaneous voiding associated with CISC.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
specific time of CISC | 1 Day
  described by the timed duration from the moment when the circumstances of care are combined to carry it out : isolated place, nearby equipment.

SECONDARY OUTCOMES:
total time of CISC | 1 Day
  described by the timed duration from the moment of the intention to self-catheter until the return to the initial activity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuro-Urology, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leroux C, Turmel N, Chesnel C, Grasland M, Le Breton F, Amarenco G, Hentzen C. Determinants and impact of the time to perform clean intermittent self-catheterization on patient adherence and quality of life: A prospective observational study. Neurourol Urodyn. 2021 Apr;40(4):1027-1034. doi: 10.1002/nau.24662. Epub 2021 Mar 26. PMID 33769589